CLINICAL TRIAL: NCT01557660
Title: Inhaled Treprostinil in Subjects With Pulmonary Arterial Hypertension: An Open-Label, Phase III, International, Multi-Center Study
Brief Title: Inhaled Treprostinil for PAH: Open-label Extension
Acronym: INTREPID - OL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PH-303
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled treprostinil (Experimental)
  Interventions: Drug: inhaled treprostinil

INTERVENTIONS:
Drug: inhaled treprostinil — 0.6mg/mL inhalation solution, up to 12 breaths four times a day

SUMMARY:
Open-label extension of RIN-PH-302.

ELIGIBILITY:
Participation and completion of all required visits for study RIN-PH-302.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Long term safety of inhaled treprostinil | up to 5 years

SECONDARY OUTCOMES:
Six-minute walk distance | up to 5 years